CLINICAL TRIAL: NCT00000483
Title: Coronary Drug Project Mortality Surveillance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 2; R01HL008888-14S1 (Other Grant/Funding Number: US NIH Grant Number)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2004-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Infarction; Myocardial Ischemia | interventions — Estrogens; Clofibrate; Dextrothyroxine; Niacin

INTERVENTIONS:
Drug: estrogen
Drug: clofibrate
Drug: dextrothyroxine sodium
Drug: niacin

SUMMARY:
To determine whether there were any long term sequelae of the drugs used in the Coronary Drug Project (estrogens, dextrothyroxine, nicotinic acid, clofibrate).

DETAILED DESCRIPTION:
BACKGROUND:

Three of the CDP treatments (two doses of estrogen and dextrothyroxine) were stopped prematurely because of toxicity. At the time the treatments were stopped, it was thought that future assessment of the status of patients on those treatments would be important to evaluate long-term sequellae. Another clinical trial evaluating clofibrate for primary prevention found that more patients on that treatment than on placebo had died. This effect persisted even after the treatment was stopped. Therefore, it was considered necessary to follow the CDP patients on clofibrate.

Of the original 834l patients, about 6000 were still alive in March l975. Cause-specific mortality in those patients was assessed through March l980.

DESIGN NARRATIVE:

The vital status of the subjects known to be alive at the end of the CDP in March l975 was assessed as of March l980. This was accomplished through questioning the local investigators, letters to the subjects, and by use of Social Security Administration and National Death Index records.

The study completion date listed in this record was obtained from the Query/View/Report (QVR) System.

ELIGIBILITY:
No eligibility criteria

Ages: 30 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1981-06; Study Completion 1985-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Sherwin — University of Maryland

REFERENCES:
- [Background] Canner PL, Klimt CR. The Coronary Drug Project. Experimental design features. Control Clin Trials. 1983 Dec;4(4):313-32. doi: 10.1016/0197-2456(83)90019-3. No abstract available. PMID 6675887
- [Background] Canner PL, Stamler J. The Coronary Drug Project. Organizational structure of the study. Control Clin Trials. 1983 Dec;4(4):333-43. doi: 10.1016/0197-2456(83)90020-x. No abstract available. PMID 6675888
- [Background] Canner PL, Berge KG, Wenger NK, Stamler J, Friedman L, Prineas RJ, Friedewald W. Fifteen year mortality in Coronary Drug Project patients: long-term benefit with niacin. J Am Coll Cardiol. 1986 Dec;8(6):1245-55. doi: 10.1016/s0735-1097(86)80293-5. PMID 3782631
- [Background] Berge KG, Canner PL. Coronary drug project: experience with niacin. Coronary Drug Project Research Group. Eur J Clin Pharmacol. 1991;40 Suppl 1:S49-51. PMID 2044644